CLINICAL TRIAL: NCT00937898
Title: BOLD (Beef in an Optimal Lean Diet) Effects on Established and Emerging Cardiovascular Disease (CVD) Risk Factors
Brief Title: Beef in an Optimal Lean Diet (BOLD) Effects on Cardiovascular Disease (CVD) Risk
Acronym: BOLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PKE101
Record Dates: First submitted 2009-06-18; First posted 2009-07-13 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Hypercholesterolemia; Hypertriglyceridemia
Keywords: lean beef; cholesterol; lipids; diet intervention
MeSH Terms: conditions — Hypercholesterolemia; Hypertriglyceridemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DASH Diet (Experimental): High fruit and vegetable, low sodium diet
  Interventions: Dietary Supplement: BOLD+ Diet; Dietary Supplement: BOLD diet
- Average American Diet (Active Comparator): Typical American diet (16% protein, ~50% carbohydrate, 33% fat)
  Interventions: Dietary Supplement: BOLD+ Diet; Dietary Supplement: BOLD diet

INTERVENTIONS:
Dietary Supplement: BOLD+ Diet — Comparison of lean beef based, high protein diet to DASH diet and Average American diet on cardiovascular disease risk factors
Dietary Supplement: BOLD diet — Comparison of lean beef based diet to DASH diet and Average American diet on risk factors of cardiovascular disease

SUMMARY:
The study is designed to assess the effects of a heart-healthy diet that includes lean beef as the primary source of high quality protein on risk factors for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. BMI > 20 and < 37
2. LDL-C level between the 50th and 90th percentile (±5% for assay variation) according to NHANES data for sex and age (ex. for men: 128-177 mg/dL and for women: 121-172 mg/dL)
3. TG level < 150 mg/dL

Exclusion criteria include:

1. self-reported history of myocardial infarction, stroke, diabetes mellitus, liver disease, kidney disease, and thyroid disease (unless controlled on medication)
2. high alcohol consumption (≥ 14 drinks/week)
3. intake of putative cholesterol-lowering supplements (psyllium, fish oil capsules, soy lecithin, niacin, fiber, flax, and phytoestrogens, stanol/sterol supplemented foods)
4. treatment with lipid-lowering agents (statins and fibrates) or blood pressure control medications
5. vegetarian diet
6. weight loss or gain ≥ 10% body weight in the previous 6 months,
7. lactation, pregnancy, or desire to become pregnant during the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-08; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Lipids (Total cholesterol, LDL-C, HDL-C, TG) | End of each 5 week diet period (weeks 5, 11, 17, 23)

SECONDARY OUTCOMES:
Apolipoprotein levels | End of each 5 week diet period (weeks 5, 11, 17, 23)
Vascular function | End of each 5 week diet period (weeks 5, 11, 17, 23)
Oxidative Stress | End of each 5 week diet period (weeks 5, 11, 17, 23)

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, Principal Investigator — Penn State University

REFERENCES:
- [Derived] Roussell MA, Hill AM, Gaugler TL, West SG, Heuvel JP, Alaupovic P, Gillies PJ, Kris-Etherton PM. Beef in an Optimal Lean Diet study: effects on lipids, lipoproteins, and apolipoproteins. Am J Clin Nutr. 2012 Jan;95(1):9-16. doi: 10.3945/ajcn.111.016261. Epub 2011 Dec 14. PMID 22170364